CLINICAL TRIAL: NCT02516904
Title: A Phase 1, Randomized, Double-Blind, Single-Dose, Dose Escalation Study to Determine the Safety, Tolerability, and Pharmacokinetics of CD101 Injection in Healthy Subjects
Brief Title: A Single Ascending Dose Study of CD101 IV in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cidara Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD101.IV.1.01
Record Dates: First submitted 2015-07-31; First posted 2015-08-06 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: Subjects
MeSH Terms: interventions — echinocandin CD101 IV

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD101 IV (Experimental): single intravenous infusion ascending dose
  Interventions: Drug: CD101 IV
- Placebo (Placebo Comparator): normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CD101 IV — antifungal
  Arms: CD101 IV
Drug: Placebo — normal saline
  Arms: Placebo

SUMMARY:
A single ascending dose study to evaluate the safety, tolerability, and pharmacokinetics of CD101 IV

DETAILED DESCRIPTION:
This is a Phase 1, single-center, prospective, randomized, double-blind study of ascending single doses of CD101 Injection administered IV to healthy adult subjects. In this study, subjects in 4 cohorts of 8 subjects, each will be randomized to receive single IV doses of CD101 Injection or placebo. Dose levels of CD101 to be assessed will follow an ascending single-dose regimen.

ELIGIBILITY:
Inclusion Criteria:

* Males surgically sterilized or using contraception,
* No significant findings on physical, ECG, clinical laboratory tests,
* BMI between 18.5 - 32.0,
* Must provide informed consent

Exclusion Criteria:

* Females of child bearing potential,
* Signs and or symptoms of an acute or chronic illness,
* Use of prescription medications within 28 days,
* Use of OTC, supplements, and herbals within 14 days,
* Current smoker
* Previous participation in a clinical study within 28 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects with clinically significant adverse events (AEs) | Up to 3 weeks

SECONDARY OUTCOMES:
Pharmacokinetic Profile as measured by: maximum plasma concentration (Cmax), time to Cmax (Tmax), area under the curve (AUC), clearance (CL), volume of distribution (Vz), elimination rate constant (^z), terminal half-life (t1/2) | Up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, MD, Principal Investigator — Celerion
Locations (1):
- Celerion Inc, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No